CLINICAL TRIAL: NCT03261193
Title: QL Block for Post-cesarean Delivery Pain
Brief Title: ITM + Bupivacaine QLB vs. ITM + Sham Saline QLB for Cesarean Delivery Pain
Acronym: qlcsection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: limited resources for recruitment
Sponsor: Nicholas Schott (Other)
Responsible Party: Sponsor-Investigator, Nicholas Schott, Anesthesiologist, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO16120234
Record Dates: First submitted 2017-07-27; First posted 2017-08-24 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Pain, Postoperative
Keywords: quadratus lumborum block; post-operative pain; cesarean section pain; analgesia; nerve block
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — SLC22A18 protein, human; Sodium Chloride; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ITM + Sham QLB (Sham Comparator): Standard spinal with intrathecal morphine for surgical anesthetic with sham saline block. Saline will be administered as a quadratus lumborum block prior to cesarean section.
  Interventions: Drug: ITM + Sham QLB
- ITM + Bupivacaine QLB (Experimental): Standard spinal with intrathecal morphine for surgical anesthetic with ql block with bupivacaine local anesthetic. Interventional drug will be administered prior to cesarean section.
  Interventions: Drug: ITM + Bupivacaine QLB

INTERVENTIONS:
Drug: ITM + Sham QLB — Sham subcutaneous non-anesthetic infiltration with saline
  Other Names: Saline
  Arms: ITM + Sham QLB
Drug: ITM + Bupivacaine QLB — QL plane block with local anesthesia
  Other Names: Bupivacaine
  Arms: ITM + Bupivacaine QLB

SUMMARY:
Comparison of standard post-operative cesarean surgery pain management with regional post-op pain control.

DETAILED DESCRIPTION:
The purpose of this trial is to determine the efficacy of a postoperative analgesia strategy that incorporates quadratus lumborum block (QLB) in conjunction with a multi-modal post-cesarean analgesia strategy. The investigators hypothesize that QLB will provide superior post-cesarean analgesia compared to the current standard of care, multi-modal analgesia.

Thus, analgesia following cesarean section using QLB compared to the current standard of care alone will be further investigated. Current practice for cesarean surgical intervention consists of multi-modal analgesia (i.e., Intrathecal morphine (ITM) and scheduled post-operative non-opioid oral analgesics, with oral opioid analgesics reserved for breakthrough pain).

Investigators will measure side-effects associated with each strategy: Standard of care methods consisting of intrathecal morphine (ITM) plus scheduled non-opioid analgesics in conjunction with prn opioid analgesics for breakthrough pain will be utilized for both. The experimental treatment arm will entail standard of care in addition to QLB. The sham comparator will entail standard of care in addition to QLB with saline.

For each strategy, we will measure and model associated economic ramifications; such factors will include drug costs, procedure costs, and costs associated with length of stay and re-admissions.

The quadratus lumborum block (QLB) is similar to the transversus abdominis plane (TAP) block, but differs slightly in regards to the anatomical region where local anesthetic is injected. Since the quadratus lumborum (QL) is more posteriorly located, it theoretically confers greater safety due to enhanced visualization. The TAP block has been studied extensively for post-cesarean delivery pain, consistently showing that it is not superior to ITM for post-operative analgesia; however, it may prove to be helpful in patients with breakthrough pain despite the use of ITM, or in patients who were unable to receive ITM (e.g. general anesthesia for cesarean, contraindications to neuraxial morphine). Thus, ITM is superior to TAP alone for post-cesarean analgesia, but it is associated with a dose-dependent increased risk for opioid related side effects. In 2015, Blanco et. al. published a study specifically using the QLB for postoperative pain after cesarean delivery. In this study, they compared a true QLB to a sham QLB all in patients who did not receive ITM, and found that the QLB provided improved pain control and decreased the need for post-operative opioids. Another study in 2016 demonstrated that the QLB is superior to the TAP block in regards to decreasing post-operative pain following c-section. Unfortunately, neither study compared the QLB to ITM (part of the current gold standard for post-cesarean delivery pain, multimodal analgesia).

The gap in knowledge regarding the utility of QLB as part of a multimodal analgesic approach including ITM for cesarean section warrants further investigation. Clinicians are constantly searching for methods to provide patients with the most effective medical interventions that provide maximal benefit and minimal harm. Post-operative pain control following cesarean delivery is an area that is important to patients and to providers, and the introduction of the QLB for this purpose has the potential to improve analgesic benefit.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean planned under spinal anesthesia
* Singleton pregnancy
* American Society of Anesthesiologists (ASA) classification score of 2 (or less)
* Gestational age of at least 37 weeks
* Intention to breastfeed infant

Exclusion Criteria:

* Contraindications to neuraxial blockade (such as clinically relevant coagulopathy, recent anticoagulant use, patient refusal, or localized skin infection overlying the site of needle entry)
* Anatomical abnormalities contraindicating spinal or QLB placement
* Received/Conversion to general anesthesia
* Received supplemental parenteral anesthesia (sedation) for any reason (e.g. unanticipated prolonged surgical procedure)
* History of chronic pain
* History of chronic opioid use/abuse
* History of Subutex, methadone, other maintenance therapy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 21 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Monroe, Study Director — University of Pittsburgh
Locations (1):
- Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.80 (4.16) | 33.35 (5.17) | 32.55 (4.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Caucasian (not Hispanic or Latino) | 10 | 11 | 21
  Black or African American (not Hispanic or Latino) | 4 | 2 | 6
  Hispanic or Latino | 0 | 0 | 0
  Asian (not Hispanic or Latino) | 1 | 0 | 1
  American Indian / Alaskan Native (not Hispanic or Latino) | 0 | 0 | 0
  Declined to answer | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29
Gravidity [Mean (Standard Deviation); unit: Number of pregnancies] | 2.93 (1.67) | 2.64 (1.08) | 2.79 (1.40)
Parity [Mean (Standard Deviation); unit: Number of births] — Number of births with a gestational age of 24 weeks or more
  Number of births | 1.27 (0.80) | 0.93 (0.47) | 1.10 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS) Pain Score With Movement
Description: Post-operative pain accompanied with patient movement will be measured using a 10-point pain scale (VAS). The VAS scale is measured with 0=no pain at all and 10=most severe pain possible.
Time Frame: 24 hours after surgical procedure (cesarean delivery)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Units on a scale | 4.85 (2.23) | 3.14 (1.83)

2. Secondary Outcome: Breast Feeding Success/Quality
Description: Limited breastfeeding resulting from pain or opioid side effects
Time Frame: 24-hours post-operatively
Population: This data was not collected during the duration of this study.
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score at Rest
Description: VAS pain score reported by the patient at rest post-operatively using a 10-point pain scale (VAS). The VAS scale is measured with 0=no pain at all and 10=most severe pain possible.
Time Frame: 1 hour after intervention
Population: Data was not collected at the specified timepoint for this outcome.
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: First Request for Pain Medication
Description: Time to first opioid dose (measured in hours)
Time Frame: From post-operative until the patient is either withdrawn from the study or requests analgesic medication up until 72 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Hours | 17.30 (14.90) | 17.37 (14.29)

5. Secondary Outcome: Sedation
Description: Presence or absence will be noted. Will be measured via Ramsay Sedation Score which ranges on a scale of 1 to 6 as follows: 1-patient is anxious, agitated, or restless. 2-patient is co-operative and oriented. 3-patient responds to commands only. 4-patient exhibits brisk response to light stimuli or loud auditory stimuli. 5-patient exhibits sluggish response to light or auditory stimuli. 6-patient exhibits no response.
Time Frame: 24-hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Participants
  Score 1 | 0 | 0
  Score 2 | 10 | 11
  Score 3 | 0 | 0
  Score 4 | 0 | 0
  Score 5 | 0 | 0
  Score 6 | 0 | 0

6. Secondary Outcome: Pruritis
Description: Presence or absence will be noted via standard pruritus scale (0-3). 0 being no evidence of pruritus, group 1 being pruritus on diseased skin, group 2 being pruritus on non-diseased skin, and group 3 being chronic reactive lesions acquired from skin manipulation, such as rubbing, picking, or scratching
Time Frame: 4-hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Participants
  Group 0 | 4 | 3
  Group 1 | 2 | 5
  Group 2 | 3 | 2
  Group 3 | 1 | 1

7. Secondary Outcome: Nausea/Vomiting
Description: Presence or absence will be noted via a scale of 0-3 as follows: 0-no nausea, 1-mild nausea not requesting pharmacological rescue, 2-moderate nausea requesting pharmacological rescue, and 3-severe nausea resistant to pharmacological treatment
Time Frame: 4-hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Participants
  Score 0 | 6 | 10
  Score 1 | 2 | 0
  Score 2 | 2 | 1
  Score 3 | 0 | 0

8. Secondary Outcome: Systolic Blood Pressure
Description: Will be measured in mmHG per standard of care and documented by study staff.
Time Frame: 4-hours post-operative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
mmHg | 113.69 (12.94) | 116.21 (12.05)

9. Secondary Outcome: Respiratory Rate
Description: Will be measured in rate/min per standard of care and documented by study staff
Time Frame: 4-hours post-operative
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Breaths/minute | 16.54 (1.76) | 16.07 (1.27)

10. Secondary Outcome: Oxygen Saturation
Description: Will be measured in % per standard of care and documented by study staff
Time Frame: 4-hours post-operative
Measure: Mean (Standard Deviation); unit: percentage of SpO2
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
percentage of SpO2 | 96.6 (2.07) | 98.4 (2.07)

11. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score at Rest
Description: as for outcome 3
Time Frame: 4 hours after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
units on a scale | 3.5 (2.77) | 1.36 (1.65)

12. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score at Rest
Description: as for outcome 3
Time Frame: 24 hours after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
units on a scale | 3.14 (1.83) | 2.38 (2.14)

13. Secondary Outcome: Visual Analogue Scale (VAS) Pain Score at Rest
Description: as for outcome 3
Time Frame: 48 hours after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
units on a scale | 3.73 (2.57) | 3.4 (2.63)

14. Secondary Outcome: Pruritis
Description: as for outcome 6
Time Frame: 24-hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Participants
  Group 0 | 5 | 5
  Group 1 | 2 | 3
  Group 2 | 2 | 2
  Group 3 | 1 | 1

15. Secondary Outcome: Pruritis
Description: as for outcome 6
Time Frame: 48-hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Participants
  Group 0 | 8 | 10
  Group 1 | 1 | 0
  Group 2 | 1 | 1
  Group 3 | 0 | 0

16. Secondary Outcome: Nausea/Vomiting
Description: as for outcome 7
Time Frame: 24-hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Participants
  Score 0 | 9 | 10
  Score 1 | 1 | 0
  Score 2 | 0 | 1
  Score 3 | 0 | 0

17. Secondary Outcome: Nausea/Vomiting
Description: as for outcome 7
Time Frame: 48-hours post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Participants
  Score 0 | 8 | 11
  Score 1 | 2 | 0
  Score 2 | 0 | 0
  Score 3 | 0 | 0

18. Secondary Outcome: Heart Rate
Description: Standard heart rate obtained
Time Frame: 4-hours post-operative
Measure: Mean (Standard Deviation); unit: Heartbeats/minute
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Heartbeats/minute | 82.62 (10.63) | 78.86 (15.94)

19. Secondary Outcome: Heart Rate
Description: Standard heart rate obtained
Time Frame: 24-hours post-operative
Measure: Mean (Standard Deviation); unit: Heartbeats/minute
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Heartbeats/minute | 86.86 (10.24) | 91.33 (6.15)

20. Secondary Outcome: Heart Rate
Description: Standard heart rate obtained
Time Frame: 48-hours post-operative
Measure: Mean (Standard Deviation); unit: Heartbeats/minute
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Heartbeats/minute | 87.00 (7.55) | 86.50 (3.54)

21. Secondary Outcome: Systolic Blood Pressure
Description: Will be measured in mmHG per standard of care and documented by study staff.
Time Frame: 24-hours post-operative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
mmHg | 109.29 (9.41) | 111.00 (11.40)

22. Secondary Outcome: Systolic Blood Pressure
Description: Will be measured in mmHG per standard of care and documented by study staff.
Time Frame: 48-hours post-operative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
mmHg | 117.6 (13.15) | 124.00 (5.66)

23. Secondary Outcome: Diastolic Blood Pressure
Description: Will be measured in mmHG per standard of care and documented by study staff.
Time Frame: 4-hours post-operative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
mmHg | 71.15 (9.21) | 70.36 (2.29)

24. Secondary Outcome: Diastolic Blood Pressure
Description: Will be measured in mmHG per standard of care and documented by study staff.
Time Frame: 24-hours post-operative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
mmHg | 68.00 (7.96) | 70.67 (8.96)

25. Secondary Outcome: Diastolic Blood Pressure
Description: Will be measured in mmHG per standard of care and documented by study staff.
Time Frame: 48-hours post-operative
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
mmHg | 75.80 (9.09) | 76.50 (7.78)

26. Secondary Outcome: Respiratory Rate
Description: Will be measured in rate/min per standard of care and documented by study staff
Time Frame: 24-hours post-operative
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Breaths/minute | 16.29 (2.93) | 16.67 (1.51)

27. Secondary Outcome: Respiratory Rate
Description: Will be measured in rate/min per standard of care and documented by study staff
Time Frame: 48-hours post-operative
Measure: Mean (Standard Deviation); unit: Breaths/minute
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
Number analyzed (Participants) | 10 | 11
Breaths/minute | 16.40 (2.19) | 18.00 (0.00)

ADVERSE EVENTS:
Time Frame: Time of consent up to 48-hours post-operative
Arm/Group | ITM + Sham QLB | ITM + Bupivacaine QLB
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT03261193/Prot_003.pdf
  • Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT03261193/SAP_004.pdf
  • Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT03261193/ICF_005.pdf